CLINICAL TRIAL: NCT02640339
Title: Retinal Abnormalities as Biomarker of Disease Progression and Early Diagnosis of Parkinson Disease
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Other Study IDs: 15-01391
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Parkinson Disease; Multiple System Atrophy; REM Sleep Behavior Disorder; Pure Autonomic Failure; Dementia With Lewy Bodies
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; REM Sleep Behavior Disorder; Pure Autonomic Failure; Lewy Body Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Parkinson Disease: Parkinson's disease is a progressive disorder of the nervous system that affects movement. It develops gradually, with alpha-synuclein deposits in neurons which aggregate into Lewy bodies.
- Mutiple system atrophy: is a degenerative neurological disorder. MSA is associated with the degeneration of nerve cells in specific areas of the brain. This cell degeneration causes problems with movement, balance, and autonomic functions of the body such as bladder control or blood-pressure regulation. Neuronal death probably occurs as a consequence of alpha-synuclein aggregation in oligodendroglia.
- REM sleep behavior disorder: a sleep disorder in which you physically act out vivid, often unpleasant dreams with vocal sounds and sudden, often violent arm and leg movements
- dementia with Lewy bodies: causes a progressive decline in mental abilities.
  It may also cause visual hallucinations, which generally take the form of objects, people or animals that aren't there. This can lead to unusual behavior such as having conversations with deceased loved ones.
  Another indicator of Lewy body dementia may be significant fluctuations in alertness and attention, which may include daytime drowsiness or periods of staring into space. And, like Parkinson's disease, Lewy body dementia can result in rigid muscles, slowed movement and tremors.
- Pure autonomic failure: Pure autonomic failure is dysfunction of many of the processes controlled by the autonomic nervous system, such as control of blood pressure•Blood pressure may decrease when people stand, and they may sweat less and may have eye problems, retain urine, become constipated, or lose control of bowel movements
- Healthy controls: Healthy normals with no neurological involvement

SUMMARY:
* To determine whether retinal abnormalities, as measured by high definition optical coherence tomography (HD-OCT) and visual electrophysiology techniques can be used as a clinical biomarker to monitor disease progression overtime in patients with Parkinson disease.
* To establish whether these measures can be used to identify patients with PD in the premotor phase.
* To define the rate of progression of retinal abnormalities in PD (both in the motor and premotor stages) for potential use as a clinical outcome measure

DETAILED DESCRIPTION:
The retina is actually brain tissue and is considered part of the central nervous system (CNS). It is the only part of the CNS that can be visualized directly and non-invasively. There is already a body of evidence that retinal neurons accumulate alpha-synuclein and degenerate in Parkinson disease (PD). Whether retinal imaging could be useful as an objective biomarker to track disease progression and response to disease-modifying treatments in patients with PD is not known.

While there are a variety of imaging techniques available (e.g., PET, SPECT, MRI), none of them has emerged as a fully reliable method to accurately measure clinical progression in PD.

The structure of the retina can be studied easily in vivo using spectral domain high definition optical coherence tomography (OCT), a non-invasive imaging technique with a resolution of ~1 microns (0.001 mm). OCT quantifies the thickness of the different retinal layers. The primary aim of this proposal is to determine whether OCT is a reliable clinical measure that can objectively measure clinical progression in PD.

Our group has shown recently that OCT can be used as a means to measure progressive neuronal loss in the retina in patients with a synucleinopathy closely related to PD (multiple system atrophy, MSA). In MSA, retinal degeneration was closely associated with disease severity and progressively worsened overtime in a predictable fashion, sufficient for biostatistical modeling. We now want to find out if this is also true in PD.

There is a panel of non-motor clinical features that increase the risk of developing PD. We propose to measure retinal nerve fiber density in these patients considering them as "pre-motor" PD and follow their clinical evolution overtime. If OCT proves useful as a means to identify pre-motor PD, such a result would present an important therapeutic window to intervene with disease modifying drugs and to prevent the development of CNS deficits.

We plan to determine whether retinal morphology can be correlated with visual function using complementary measures of visual electrophysiology techniques, including pattern electroretinogram (PERG) and photopic negative response (PhNR). These techniques have been used in patients with PD and other synucleinopathies, and do map closely to retinal function abnormalities. But, there is little data describing how these functional measure of the retina progression over time in PD.

We hypothesize that patients with PD have specific patterns of damage in retinal structure and function, that this pattern can be identified in the premotor phase, We believe that OCT can be used as an objective biomarker of premotor diagnosis and disease progression.

INNOVATION:

The structure of the retina presents an ideal opportunity to image the CNS overtime with OCT. As a widely available clinical technique that correlates closely with functional measures of visual electrophysiology, OCT is being increasingly used in multiple sclerosis and other neurodegenerative disorders. If successful, this work may provide a significant tool for the diagnosis of PD in the pre-motor phase and could be used as a clinical outcome measure in disease-modifying trials. To achieve these objectives, we will take advantage of the infrastructure used in the ongoing NIH-funded Natural History of Autonomic Disorders study (ClnicalTrials.gov: NCT01799915), which prospectively follows patients with synucleinopathies with standardized neurological measures overtime. The proposal will provide measures of retinal structure in conjunction with measures of disease severity in a group of patients with well-defined PD. By measuring retinal structure in a group of patients considered high risk for developing PD (namely REM sleep behavior disorder -RBD, and isolated autonomic failure) we will determine the usefulness of OCT as a mean to identify PD in the premotor phase.

ELIGIBILITY:
Inclusion Criteria:

Subjects with PD, MSA and DLB that fulfill current diagnostic criteria.

* Subjects with RBD that have polysomnography-confirmed diagnosis showing evidence of lack of muscle atonia and dream enacting behaviors during REM sleep.
* Subjects with isolated autonomic failure (i.e., no motor deficits) that have evidence of neurogenic orthostatic hypotension and other features of autonomic failure without clinical evidence of cognitive impairment.
* Control subjects with no history of neurological or ophthalmological disorders.

Exclusion Criteria:

* Subjects with glaucoma, retinopathy, or significant media opacification (e.g., cataracts).
* Subjects with a history of eye surgery or eye trauma
* Inability to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will select patients from our clinic and take advantage of the infrastructure used in the ongoing NIH-funded Natural History of Autonomic Disorders study (ClnicalTrials.gov: NCT01799915), which prospectively follows patients with synucleinopathies with standardized neurological measures overtime.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2016-02; Primary Completion 2020-09 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Retinal nerve fiber layer (RNFL) thickness | Every 6 months from baseline to 3 years
  The results of the RNFL thickness will be expressed in microns in different zones around the optic nerve: temporal, superior, nasal, inferior and global.
Retinal ganglion cell layer (GCL) thickness | Every 6 months from baseline to 3 years
  The results of the GCL thickness will be expressed in microns in different zones around the fovea region: temporal- superior, superior, nasal-superior, nasal inferior, inferior, temporal inferior and global.

SECONDARY OUTCOMES:
• Visual Acuity | Every 6 months from baseline to 3 years
  Will be expressed in decimal units
• Color Discrimination | Every 6 months from baseline to 3 years
  Will be expressed in decimal units.
• Pupillometry | Every 6 months from baseline to 3 years
  Measures will include pupil diameter (expressed in millimeters, in dark and light conditions and the amplitude and velocity of the pupillary response.
• Videonystagmography | Every 6 months from baseline to 3 years
  Saccadic velocity and amplitude (expressed in m/seg and degrees) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Horacio C Kaufmann, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No